CLINICAL TRIAL: NCT00005912
Title: An Open Intravenous Multiple Dose, Multi-Center Study to Investigate the Pharmacokinetics, Safety and Toleration of Voriconazole in Children Aged 2-12 Years Who Require Treatment for the Prevention of Systemic Fungal Infection
Brief Title: Voriconazole to Prevent Systemic Fungal Infections in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000150; 00-C-0150
Record Dates: First submitted 2000-06-14; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-06

CONDITIONS: Aspergillosis; Candidiasis; Fungal Diseases; Mycoses
Keywords: Aspergillosis; Candidiasis; Fungal Infections; Fungemia; Prophylactic Antifungal Therapy; Pediatric Fungal Infection
MeSH Terms: conditions — Aspergillosis; Candidiasis; Mycoses; Fungemia | interventions — Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
This study will examine how children's bodies metabolize and eliminate the anti-fungal drug voriconazole. The results will yield information needed to make recommendations for safe and effective dosing of the drug in children. Children with reduced immune function-such as those receiving drugs for cancer treatment-are at high risk for serious fungal infections.

Children between 2 and 12 years old who need treatment to prevent fungal infections may be eligible for this study. Candidates will be screened with a physical examination, eye examination, and blood and urine tests.

Children in the study will be hospitalized for 21 days. They will receive voriconazole twice a day (every 12 hours) for 8 days, infused through a vein over a period of 1 to 2 hours. The dose will be determined based on the individual child's weight. Blood samples will be collected at various intervals before and after the infusions on days 1, 2, 4 and 8 to determine the amount of drug in the blood. On day 8, the child will have another physical and eye examination, as well as additional blood and urine tests. If additional treatment is required, voriconazole may be continued for up to day 21. (Children who require the drug for more than 21 days may receive it under another research protocol.) On the last day of treatment, the child will have another physical examination, and blood and urine tests. These procedures will be repeated again at 30 to 35 days following the last dose of drug. A small sample of blood will also be analyzed for genetic information related to the rate of metabolism of voriconazole-that is, how fast or slow it is cleared (eliminated) by the liver.

Voriconazole is effective against several different fungi. It may protect children against serious fungal infections with fewer side effects than standard available therapy.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the serum levels and pharmacokinetic parameters achieved following two dosage levels of voriconazole. In addition, the safety and toleration of intravenous voriconazole at two dosage levels in an immunocompromised pediatric patient population will be evaluated. Also, the plasma concentrations of the major metabolite of voriconazole (N-oxide) in these patients will be performed. The study is designed as a multi-center, open label multi-dose study of intravenous voriconazole. Intravenous voriconazole will be administered prophylactically twice daily to immunocompromised children at high risk for invasive mycoses. The patient population consists of children ages 2 years to 12 years of age; two age groups will be studied (2-<6, 6-12). Initial dosage levels will be 3mg/kg q12h and 4mg/kg q12h. The planned sample size is 24 children. For those children who do not complete the full 8 days of kinetics, a replacement patient will be added. Immunocompromised children at high risk for invasive mycoses will receive voriconazole prophylactically. Therapy will be initiated within 48 hours after completion of chemotherapy. Voriconazole therapy will continue until recovery from neutropenia. The first 12 children will initially receive a loading dose of 6mg/kg X 2 doses followed by 3mg/kg BID through day 4 of therapy. Twelve hour pharmacokinetics will be collected on day 4. Children will then receive 4mg/kg starting on the second dose of day 4 and will continue at that dosage level until recovery from neutropenia. Kinetics will again be collected at the 4mg/kg dosage level on day 8 of therapy. If the mean peak plasma concentration of voriconazole in the first 12 patients following 4mg/kg q12h dosing is less than 4,000ng/ml., the remaining 12 patients will receive voriconazole after day 4 at a dosage of 5mg/kg.

ELIGIBILITY:
Children (male or female) ages 2-12 years who require treatment for the prevention of systemic fungal infection.

Children who are expected to develop neutropenia lasting for more than 10 days following chemotherapy for one of the following conditions: leukemia, lymphoma, aplastic anemia, or as the preparative regimen for bone marrow transplantation.

Patients who are anticipated to live more than 3 months.

Females of child-bearing potential (post-menarchal) must have a negative pregnancy test at entry.

Informed consent of the parent or legally authorized representative obtained prior to entry.

Assent will be obtained from minors capable of understanding.

No patients who are receiving and cannot discontinue the following drugs at least 24 hours prior to study start: terfenadine and cisapride (due to the possibility of QTc prolongation). Omegprazole (an inhibitor of CYP2C19) which is known to increase plasma voriconazole levels.

No patients who have received the following drugs within 14 days prior to study entry: rifampicin, rifabutin, carbamazepine, phenytoin, nevirapine and barbiturates as these are potent inducers of hepatic enzymes and will result in undetectable levels of voriconazole.

No patients who have received astemizole within the previous 60 days.

No patients who are taking or are likely to receive any investigational drugs except: used for cancer treatment, antiretroviral agents, and drugs used for treatments of any AIDS defining opportunistic infections.

No patients with a history or hypersensitivity to or severe intolerance of azole antifungal agents.

No patients who have already been entered onto this protocol once.

No patient with medical history or evidence of cardiac arrhythmia.

No patients with AST and ALT greater than or equal to 5XULN.

No patients with moderate and severe renal impairment (i.e., calculated creatine clearance less than 30ml/min). If creatinine clearance is reduced to less than 30 ml/min at any time during the study, the patient must be discontinued from the study. Creatine clearance will be calculated using the following equation: 0.55 X height (cm)/serum creatinine (mg/dL).

Any other condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 2000-06; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Walsh TJ, Hiemenz JW, Anaissie E. Recent progress and current problems in treatment of invasive fungal infections in neutropenic patients. Infect Dis Clin North Am. 1996 Jun;10(2):365-400. doi: 10.1016/s0891-5520(05)70303-2. PMID 8803625
- [Background] Pizzo PA, Robichaud KJ, Gill FA, Witebsky FG. Empiric antibiotic and antifungal therapy for cancer patients with prolonged fever and granulocytopenia. Am J Med. 1982 Jan;72(1):101-11. doi: 10.1016/0002-9343(82)90594-0. No abstract available. PMID 7058815
- [Background] Walsh TJ, Gonzalez C, Lyman CA, Chanock SJ, Pizzo PA. Invasive fungal infections in children: recent advances in diagnosis and treatment. Adv Pediatr Infect Dis. 1996;11:187-290. No abstract available. PMID 8718464